CLINICAL TRIAL: NCT05364021
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-escalation Study to Investigate the Safety, Tolerability, PK, PD, and Exploratory Efficacy of LP352 in Subjects With Developmental and Epileptic Encephalopathies
Brief Title: Study to Investigate LP352 in Subjects With Developmental and Epileptic Encephalopathies
Acronym: PACIFIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Longboard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP352-201
Record Dates: First submitted 2022-03-22; First posted 2022-05-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Developmental and Epileptic Encephalopathy; Dravet Syndrome; Lennox Gastaut Syndrome
Keywords: CDKL5 deficiency disorder; developmental and epileptic encephalopathy; Dravet Syndrome; epilepsy; Lennox-Gastaut Syndrome; treatment resistant epilepsy; tuberous sclerosis complex
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome; CDKL5 deficiency disorder; Epilepsy; Tuberous Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LP352 (Experimental): Subjects will be titrated up to highest tolerated dose of LP352 during a 15-day period, followed by a 60-day maintenance period and a 15-day taper/down titration period.
  Interventions: Drug: LP352
- Placebo (Placebo Comparator): Placebo for LP352
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LP352 — LP352 administered three times daily, orally or through G-tube
  Arms: LP352
Drug: Placebo — Matching placebo for LP352 administered three times daily, orally or through G-tube
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety, tolerability, efficacy, and pharmacokinetics of adjunctive therapy of LP352 in adults and adolescents with developmental and epileptic encephalopathies.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, dose-escalation, placebo-controlled study of LP352 in adults and adolescents with developmental and epileptic encephalopathies (DEE) with an average of ≥ 4 observed/countable motor seizures per 4-week period during the 12 weeks before screening while on stable antiseizure medicine (ASM).

Subjects will be randomized 4:1 to LP352 or placebo. The study will have a baseline period of 28 days, followed by a 15 day up-titration period during which time subjects will titrate up to their highest tolerated doses, and a 60-day maintenance period. After Day 75, subjects will be tapered down over a period of up to 15 days, with a follow-up visit 30 days after last dose. Enrolled subjects will be allowed to continue treatment with up to 4 concomitant ASMs at a stable dose.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, age 12 to 65 years
2. Diagnosis of Dravet syndrome, Lennox-Gastaut syndrome, or other developmental and epileptic encephalopathy
3. Has a minimum number of seizures per 4-week period while taking 1 to 4 anti-seizure medications
4. All medications and epilepsy interventions must be stable for 4 weeks before screening and are expected to remain stable during the study
5. The patient/parent/caregiver is able and willing to attend study visits, complete the diary and take study drug as instructed

Key Exclusion Criteria:

1. Current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, pulmonary arterial hypertension or abnormal blood pressure
2. Has glaucoma, renal impairment, liver disease or any other medical condition that would affect study participation or pose a risk to the subject
3. Current or recent history of moderate or severe depression, anorexia nervosa, bulimia or at risk of suicidal behavior
4. Currently taking anorectic agents, monoamine oxidase inhibitors; serotonin agonists or antagonists including fenfluramine, atomoxetine, vortioxetine, or other medications for weight loss
5. Positive test result on the drug screen, except tetrahydrocannabinol (THC) for patients taking prescribed cannabidiol

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events | Baseline up to Day 75
  Incidence and severity of adverse events, including serious adverse events and adverse events leading to study discontinuation and clinically significant changes in vital signs, physical examination endpoints, clinical safety laboratory values and ECGs
Columbia-Suicide Severity Rating Scale (C-SSRS) Response | Baseline up to Day 75
  Type of Suicidal Ideation, Intensity (1 - 5, with 5 being most severe), Suicidal Behavior
Patient Health Questionnaire-9 Total Score and Question 9 Score | Baseline up to Day 75
  Severity Rating Scale: 0 - 27; higher scores indicate greater severity of depressive disorder
Percent Change from Baseline in Observed Countable Motor Seizure Frequency (per 28 Days) During the Treatment Period | Baseline up to Day 75
Percent Change from Baseline in Observed Countable Motor Seizure Frequency (per 28 Days) During the Maintenance Period | Baseline up to Day 75

SECONDARY OUTCOMES:
Observed Plasma Concentrations of LP352 by Time and Dose | Baseline up to Day 75
Modeled Estimate of Average Plasma Concentration | Baseline up to Day 75
Modeled Estimate of Observed Plasma Concentration Just Prior to Dosing | Baseline up to Day 75
Correlation of Plasma Concentration with Incidence of Treatment-emergent Adverse Events | Baseline up to Day 75
Correlation of Plasma Concentration with Seizure Frequency | Baseline up to Day 75
Observed and Change from Baseline Prolactin Concentration During the Treatment Period | Baseline up to Day 75

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Dlugos, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (34):
- United States (29):
  - University of Arizona - Health Sciences Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rancho Los Amigos National Rehabilitation Center (RLANRC), Downey, California
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Northwest Florida Clinical Research Group, Gulf Breeze, Florida
  - University of Miami, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Research Institute of Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, Boise, Idaho
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Boston Children's Health Physicians LLP, Hawthorne, New York
  - New York University Langone Hospital - Long Island, Mineola, New York
  - Northwell Health, New York, New York
  - Northeast Regional Epilepsy Group, Staten Island, New York
  - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Providence Neurological Specialties-East, Portland, Oregon
  - Child Neurology Consultants of Austin, Austin, Texas
  - Austin Epilepsy Care Center, Austin, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington Valley Medical Center, Renton, Washington
- Australia (5):
  - Royal Brisbane Women's Hospital, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Children's Hospital, Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No